CLINICAL TRIAL: NCT04003207
Title: An Open Label Trial of Growth Hormone in Children and Adolescents With Phelan-McDermid Syndrome Targeting Social Withdrawal
Brief Title: Growth Hormone Treatment in Children With Phelan McDermid Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swathi Sethuram (Other)
Responsible Party: Sponsor-Investigator, Swathi Sethuram, Fellow, Division of Pediatric Endocrinology & Diabetes, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-2549
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Phelan McDermid Syndrome
Keywords: Phelan McDermid Syndrome; 22q13 deletion Syndrome; Growth hormone; Autism; Insulin like growth factor 1
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Autistic Disorder | interventions — Growth Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phelan-McDermid syndrome (Experimental): Patients with Phelan-McDermid syndrome receive 12 weeks of growth hormone therapy
  Interventions: Drug: Recombinant human Growth hormone

INTERVENTIONS:
Drug: Recombinant human Growth hormone — Subcutaneous growth hormone injections given once daily at a dose between 0.15mg/kg/week to 0.47 mg/kg/week titrated based on IGF-1 levels in serum for a duration of 12 weeks.

SUMMARY:
Phelan McDermid syndrome (PMS) is a rare genetic form of autism spectrum disorder (ASD) due to deletions or mutations in the SHANK3 gene. This is a pilot open labeled trial of growth hormone therapy in children with PMS targeting social withdrawal and repetitive behavior. This research study will include children with PMS between 2-12 years of age who will receive growth hormone daily for 12 weeks, if found to be eligible. The aim of this study is to evaluate the effect of growth hormone on behavioral outcomes such as the aberrant behavior checklist social withdrawal subscale (ABC-SW) and repetitive behavior scale- revised (RBS-R). The effects of growth hormone on visual evoked potentials will also be assessed. Growth hormone increases insulin like growth factor 1 (IGF-1) levels and a previous trial of IGF-1 therapy in PMS children showed improvement in these behavioral scales. Growth hormone has been studied for decades with an excellent safety profile and fewer adverse effects compared to IGF-1 therapy in other conditions. Hence, this may be a viable therapeutic option. There is no treatment currently available for PMS and this trial is therefore extremely important.

DETAILED DESCRIPTION:
BACKGROUND: Phelan-McDermid syndrome (PMS) is a genetic form of autism spectrum disorder (ASD) associated with developmental delay and hypotonia. IGF-1 promotes brain vessel growth, neurogenesis, and synaptogenesis.

The research team previous clinical trial of IGF-1 in patients with Phelan McDermid Syndrome has shown improvement in core ASD symptoms using the Aberrant Behavior Checklist (ABC) and the Repetitive Behavior Scale-Revised (RBS-R). Growth hormone (GH) binds to its receptor and initiates a cascade of events which directly increases synthesis and release of IGF-1 levels. HYPOTHESIS: The study team hypothesize that rise in IGF-1 stimulated by growth hormone (GH) administration should produce improvement in behavior in children and adolescents with PMS as previously demonstrated with use of IGF-1.

RESEARCH PLAN: The study team seek to recruit 10 patients with PMS and administer growth hormone as once daily subcutaneous injections for 12 weeks at standard doses. The study team will monitor baseline anthropometric measures, laboratory parameters for growth, IGF-1 levels, and bone age prior to therapy and continue to monitor safety laboratory parameters during and after therapy. The goal of therapy would be to maintain IGF-1 levels between 1-2SD above the mean for age and puberty. Evaluations will include validated behavioral scales. Visual evoked potentials (VEPs) will be used as biomarkers of visual sensory reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Known pathogenic deletions or mutations in SHANK3 gene diagnosed by array CGH and/or direct sequencing.
* Children between 2 and 12 years of age.
* Open epiphyses on bone age x ray

Exclusion Criteria:

* closed epiphyses;
* active or suspected neoplasia;
* intracranial hypertension;
* hepatic insufficiency;
* renal insufficiency;
* cardiomegaly/valvulopathy;
* history of allergy to growth hormone or any component of the formulation (mecasermin);
* history of extreme prematurity (<1000 grams) with associated early neo-natal complications, e.g. intra-cerebral
* hemorrhage, prolonged hypoxia, prolonged hypoglycemia;
* patients with comorbid conditions who are deemed too medically compromised to tolerate the risk of experimental treatment with growth hormone.
* Patient with visual problems that preclude the use of VEP's

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Sethuram, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Alexander Kolevzon, MD, Study Director — Icahn School of Medicine at Mount Sinai; Robert Rapaport, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Seaver Autism Center, New York, New York, United States

REFERENCES:
- [Background] Kolevzon A, Bush L, Wang AT, Halpern D, Frank Y, Grodberg D, Rapaport R, Tavassoli T, Chaplin W, Soorya L, Buxbaum JD. A pilot controlled trial of insulin-like growth factor-1 in children with Phelan-McDermid syndrome. Mol Autism. 2014 Dec 12;5(1):54. doi: 10.1186/2040-2392-5-54. eCollection 2014. PMID 25685306
- [Background] De Rubeis S, Siper PM, Durkin A, Weissman J, Muratet F, Halpern D, Trelles MDP, Frank Y, Lozano R, Wang AT, Holder JL Jr, Betancur C, Buxbaum JD, Kolevzon A. Delineation of the genetic and clinical spectrum of Phelan-McDermid syndrome caused by SHANK3 point mutations. Mol Autism. 2018 Apr 27;9:31. doi: 10.1186/s13229-018-0205-9. eCollection 2018. PMID 29719671
- [Background] Costales J, Kolevzon A. The therapeutic potential of insulin-like growth factor-1 in central nervous system disorders. Neurosci Biobehav Rev. 2016 Apr;63:207-22. doi: 10.1016/j.neubiorev.2016.01.001. Epub 2016 Jan 15. PMID 26780584
- [Background] Grimberg A, DiVall SA, Polychronakos C, Allen DB, Cohen LE, Quintos JB, Rossi WC, Feudtner C, Murad MH; Drug and Therapeutics Committee and Ethics Committee of the Pediatric Endocrine Society. Guidelines for Growth Hormone and Insulin-Like Growth Factor-I Treatment in Children and Adolescents: Growth Hormone Deficiency, Idiopathic Short Stature, and Primary Insulin-Like Growth Factor-I Deficiency. Horm Res Paediatr. 2016;86(6):361-397. doi: 10.1159/000452150. Epub 2016 Nov 25. PMID 27884013
- [Background] Aramburo C, Alba-Betancourt C, Luna M, Harvey S. Expression and function of growth hormone in the nervous system: a brief review. Gen Comp Endocrinol. 2014 Jul 1;203:35-42. doi: 10.1016/j.ygcen.2014.04.035. Epub 2014 May 13. PMID 24837495
- [Derived] Sethuram S, Levy T, Foss-Feig J, Halpern D, Sandin S, Siper PM, Walker H, Buxbaum JD, Rapaport R, Kolevzon A. A proof-of-concept study of growth hormone in children with Phelan-McDermid syndrome. Mol Autism. 2022 Jan 29;13(1):6. doi: 10.1186/s13229-022-00485-7. PMID 35093163

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phelan-McDermid Syndrome
Started | 6
Completed | 5
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: ABC - Social Withdrawal Subscale
Description: A caregiver report symptom checklist. 58-item instrument into 5 subscales: Irritability (score 0-45); Lethargy/Social Withdrawal (score 0-48); Stereotypic Behavior (score 0-21); Hyperactivity (score 0-48); Inappropriate Speech (score 0-12). Total scale 0-174, with higher score indicating more aberrant behavior.
Time Frame: After 12 weeks of growth hormone therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 6
score on a scale
  Irritability baseline | 10.31 (7.6)
  Irritability 12 weeks | 4.6 (2.3)
  Social Withdrawal baseline | 14.8 (7.4)
  Social Withdrawal 12 weeks | 6.2 (3.4)
  Stereotypy baseline | 8.8 (6.9)
  Stereotypy 12 weeks | 5.1 (1.8)
  Hyperactivity baseline | 33.3 (6.2)
  Hyperactivity 12 weeks | 16.5 (7.7)
  Inappropriate Speech baseline | 3.3 (4.3)
  Inappropriate Speech 12 weeks | 2.3 (3.8)

2. Primary Outcome: Repetitive Behavior Scale-Revised (RBS-R)
Description: A 43 item instrument with total score from 0-129, with higher score indicating more restricted, repetitive and stereotyped behaviors.
  Subscales
  Stereotyped Behavior (0-27)
  Self-injurious Behavior (0-24)
  Compulsive Behavior (0-18)
  Ritualistic Behavior (0-36)
  Sameness Behavior (0-33)
  Restricted Behavior (0-12)
Time Frame: After 12 weeks of growth hormone therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 6
score on a scale
  Stereotyped Behavior at baseline | 4.3 (1.7)
  Stereotyped Behavior at Week 12 | 4.0 (2.4)
  Self-injurious Behavior at baseline | 0.7 (0.8)
  Self-injurious Behavior at Week 12 | 1.3 (1.8)
  Compulsive Behavior at baseline | 2.8 (3.2)
  Compulsive Behavior at Week 12 | 1.3 (1.6)
  Ritualistic Behavior at baseline | 1.2 (1.2)
  Ritualistic Behavior at Week 12 | 0.8 (1.2)
  Sameness Behavior at baseline | 2.3 (2.4)
  Sameness Behavior at Week 12 | 2.0 (1.7)
  Restricted Behavior at baseline | 2.0 (2.2)
  Restricted Behavior at Week 12 | 1.2 (1.5)
  Total at baseline | 13.3 (6.1)
  Total at Week 12 | 10.7 (3.1)

3. Primary Outcome: The Sensory Profile
Description: The full Sensory Profile has 125 items and the short version contains 38 items. Parents use a Likert scale to rate how frequently their child demonstrates a particular behavior (ranging from 1 = always to 5 = never).
  Total scale for the Short Sensory Profile 38-190, with a lower score indicates greater deviation from typically developing children and indicates more sensory reactivity symptoms.
  Subscales
  Tactile (7-35)
  Taste / Smell (4-20)
  Movement (3-15)
  Sensation (7-35)
  Auditory (6-30)
  Low Energy / Weak (6-30)
  Visual / Auditory (5-25)
Time Frame: After 12 weeks of growth hormone therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 6
score on a scale
  Tactile at Baseline | 31.5 (2.1)
  Tactile at Week 12 | 31.7 (2.0)
  Taste / Smell at Baseline | 18.2 (3.6)
  Taste / Smell at Week 12 | 19.4 (1.3)
  Movement at Baseline | 13.3 (1.6)
  Movement at Week 12 | 13.7 (1.8)
  Sensation at Baseline | 17.5 (4.8)
  Sensation at Week 12 | 20.0 (3.8)
  Auditory at Baseline | 20.0 (1.9)
  Auditory at Week 12 | 22.0 (2.4)
  Low Energy / Weak at Baseline | 16.5 (6.9)
  Low Energy / Weak at Week 12 | 20.5 (5.2)
  Visual / Auditory at Baseline | 22.3 (2.3)
  Visual / Auditory at Week 12 | 22.7 (1.5)
  Total at Baseline | 139.3 (12.7)
  Total at Week 12 | 148.8 (12.8)

4. Primary Outcome: The Sensory Assessment for Neurodevelopmental Disorders (SAND)
Description: a clinician-administered assessment and corresponding caregiver interview that is not dependent on verbal or cognitive ability and is therefore appropriate for severely affected or nonverbal individuals with PMS. Responses are rated by a trained examiner on an algorithm. Scores are dichotomous, 0 (not present) or 1 (present) and are based on a summary of observed sensory behaviors throughout the duration of the observation. A total SAND score ranging from 0 to 90. Higher scores represent a higher level of sensory reactivity symptoms.
Time Frame: After 12 weeks of growth hormone therapy
Population: Data not collected due to pandemic.
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 0

5. Secondary Outcome: Visual Evoked Potentials (VEP)
Description: A noninvasive technique to evaluate the functional integrity of visual pathways in the brain from the retina to the visual cortex via the optic nerve/optic radiations. The VEP is recorded from the head's surface, over the visual cortex, and is extracted from ongoing EEG through signal averaging. VEPs reflect the sum of excitatory and inhibitory postsynaptic potentials occurring on apical dendrites (Zemon et al., 1986) which modulate excitatory and inhibitory signals received by the pyramidal cells.
Time Frame: After 12 weeks of growth hormone therapy
Population: Data not collected due to pandemic.
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Auditory Event Related Potentials (AERP)
Description: AERP is useful for characterizing early processing of auditory tones and habituation to rapidly repeated stimuli as in speech processing. AERP amplitudes are measured at 12 weeks and compared to baseline.
Time Frame: Baseline and 12 weeks of growth hormone therapy
Population: Data not collected due to pandemic.
Arm/Group | Phelan-McDermid Syndrome
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Phelan-McDermid Syndrome
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phelan-McDermid Syndrome (N=6)
Increase in appetite (Gastrointestinal disorders) | 3
Gastroenteritis (Gastrointestinal disorders) | 3
Polyuria/nocturia (Renal and urinary disorders) | 3
Crying spells (Psychiatric disorders) | 3
Runny nose/cough/sneezing (General disorders) | 3
Decrease in appetite (Gastrointestinal disorders) | 2
Fever (Infections and infestations) | 2
Worsening repetitive behavior (Psychiatric disorders) | 2
Eye/ear infection (Infections and infestations) | 2
Diarrhea (Gastrointestinal disorders) | 1
Worsening hyperactivity (General disorders) | 1
Sleep disturbance (Psychiatric disorders) | 1
Disruptive behavior (Psychiatric disorders) | 1
Bruising at injection site (Skin and subcutaneous tissue disorders) | 1
Sweating of hands/feet (General disorders) | 1
Limping/gait changes (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04003207/Prot_SAP_000.pdf